CLINICAL TRIAL: NCT05530720
Title: Acceptance of Complementary Medicine in Germany - an Anonymous Representative Cross-sectional Study Including a Qualitative Survey
Brief Title: Acceptance of Complementary Medicine in Germany
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Otto-Friedrich-University Bamberg, Chair of Sociology, Prof. Dr. Rasmus Hoffmann (Unknown)
Responsible Party: Principal Investigator, Dr. Christian S. Kessler, Principal Investigator, Charite University, Berlin, Germany
Other Study IDs: Complementary Medicine Survey
Record Dates: First submitted 2022-08-26; First posted 2022-09-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: General Population
MeSH Terms: interventions — Cross-Sectional Studies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Online survey with 3.000 participants using mobile website technology
  Interventions: Other: Cross-sectional survey

INTERVENTIONS:
Other: Cross-sectional survey — No intervention.

SUMMARY:
Complementary medicine is widely practiced in Germany and worldwide. The aim of this study is to explore how many people use complementary medicine methods in Germany, for which health-related issues they do and for which they would not.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Age at least 18 years
* Sufficient language skills as well as cognitive ability to participate in an online survey or interview lasting approximately 30 minutes
* Active consent to the online consent form

Exclusion Criteria:

- Lack of consent to participate in the study

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Respondents are recruited from Respondi institute's pool of test persons, but remain completely anonymous with regard to their personal data and answers; they are also not subsequently or indirectly identifiable.
Sampling Method: Probability Sample
Enrollment: 4505 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2022-10-17 (Actual); Study Completion 2022-10-17 (Actual)

PRIMARY OUTCOMES:
Assessment of attitudes towards complementary medicine | Up to 24 weeks
  Assessed retrospectively with self-designed questions

SECONDARY OUTCOMES:
Sociodemographic Parameters | Up to 24 weeks
  Assessed retrospectively with self-designed questions
Assessment of knowledge of complementary medicine | Up to 24 weeks
  Assessed retrospectively with self-designed questions
Assessment of own application of complementary medicine | Up to 24 weeks
  Assessed retrospectively with self-designed questions
Assessment of medical history and quality of life by EQ-5D-5L | Up to 24 weeks
  Assessed retrospectively with self-designed questions
Assessment of attitudinal and behavioral questions (e.g. lifestyle) | Up to 24 weeks
  Assessed retrospectively with self-designed questions
Assessment of use of complementary medicine in the Covid-19 pandemic | Up to 24 weeks
  Assessed retrospectively with self-designed questions

OTHER OUTCOMES:
Qualitative interviews of experts | Conducted after completion of the questionnaire (once), up to 24 weeks
Qualitative interviews of participants | Conducted after completion of the questionnaire (once), up to 24 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Otto-Friedrich-University Bamberg, Bamberg
  - Charité Hochschulambulanz für Naturheilkunde, Immanuel Krankenhaus Berlin, Berlin

REFERENCES:
- [Derived] Ortiz M, Wischnewsky M, Jeitler M, Brinkhaus B, Michalsen A, Hoffmann R, Kessler CS. Health-Related quality of life and the impact of traditional, complementary and integrative Medicine - an Online - Representative Cross-Sectional survey in Germany. BMC Public Health. 2025 Aug 21;25(1):2870. doi: 10.1186/s12889-025-23908-5. PMID 40841634